CLINICAL TRIAL: NCT00021216
Title: A Phase I Study Of PS-341 In Pediatric Patients With Refractory Solid Tumors
Brief Title: Bortezomib in Treating Children With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01860; NCI-2012-01860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0015; CDR0000068760; ADVL0015 (Other: Children's Oncology Group); ADVL0015 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Phase I trial to study the effectiveness of bortezomib in treating children who have advanced solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib in pediatric patients with refractory solid tumors.

II. Determine the dose-limiting toxicity and other toxic effects of this regimen in these patients.

III. Preliminarily determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. If dose-limiting toxicity in the form of myelosuppression occurs in stratum I, dose escalation continues with patients meeting the qualifications for stratum II.

PROJECTED ACCRUAL: Approximately 24-36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is refractory to standard therapy or for which no standard therapy exists

  * Histologic confirmation not required for brainstem glioma or optic pathway tumor
* Ineligible for therapies of higher priority
* Stratum II only:

  * No bone marrow involvement
* Performance status - Karnofsky 50-100% (over 10 years of age)
* Performance status - Lansky 50-100% (10 years of age and under)
* At least 8 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)
* Hemoglobin at least 8 g/dL (RBC transfusions allowed)
* Bilirubin less than 1.5 mg/dL
* ALT less than 5 times normal for age
* Albumin at least 2 g/dL
* Creatinine no greater than upper limit of normal for age
* Creatinine clearance or radioisotope glomerular filtration rate greater than 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologic deficits related to CNS tumors allowed if relatively stable for at least 2 weeks
* No uncontrolled infection
* At least 7 days since prior biologic therapy and recovered
* At least 3 months since prior allogeneic stem cell transplantation
* At least 1 week since prior growth factors
* Stratum II only:

  * No prior stem cell transplantation with or without total body irradiation
* At least 2 weeks since prior chemotherapy (4 weeks for nitrosoureas) and recovered
* Stratum II only:

  * No more than 2 prior multi-agent chemotherapy regimens
  * More than 2 single-agent regimens allowed
* Concurrent dexamethasone allowed for CNS tumors if stable dose for at least 2 weeks
* See Biologic therapy
* At least 2 weeks since prior palliative local radiotherapy
* At least 6 months since prior craniospinal radiotherapy or radiotherapy to at least 50% of pelvis
* At least 6 weeks since prior substantial bone marrow radiotherapy
* Recovered from prior radiotherapy
* Stratum II only:

  * No prior radiotherapy to more than 20% of bone marrow
* No prior bortezomib
* No concurrent anticonvulsants
* No other concurrent investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2001-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose at which fewer than 20% of patients experience DLT assessed using CTC version 2.0 | 3 weeks
20S proteasome inhibition | Up to 2 weeks
  The 95% confidence interval for the percent of patients who exhibit inhibition at a recommended dose level determined according to the table above is 61%-100%, if six patients are evaluated or 55%-100% if five patients are evaluated.
Progression free survival | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States